CLINICAL TRIAL: NCT06034392
Title: CHAMP App Cardiac Study: Evaluation of Software Functions for Asynchronous Monitoring of Children With Complex Congenital Heart Disease in the Home Setting and Data Repository
Brief Title: CHAMP App Cardiac Study and Repository
Acronym: CHAMP
Status: Enrolling by invitation | Type: Observational
Sponsor: Lori Erickson (Other)
Responsible Party: Sponsor-Investigator, Lori Erickson, Director, Remote Health Solutions, Children's Mercy Hospital Kansas City
Organization: Children's Mercy Hospital Kansas City (Other)
Other Study IDs: 15030113CMH
Record Dates: First submitted 2023-08-24; First posted 2023-09-13 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Heart Defects, Congenital; Pediatrics
Keywords: mHealth; Software Platform
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: CHAMP App — CHAMP® App is a downloadable software mobile Application with a Software Platform. CHAMP® App is an electronic version of data entry for children with conditions that require close monitoring from their homes. The primary Intended Use is to relay monitoring information from homes to the health care team. This monitoring includes data options that can facilitate the collection of monitoring data of children in the home setting to improve communications between parents at home and remote caregivers. The CHAMP® App itself does not do home monitoring of the child's medical condition. It is not designed to alert parents if data entered has reached a red flag (problem) level. Users of the CHAMP App are advised in writing and in the informed consent process that urgent medical conditions should not be managed through the CHAMP App, and that appropriate emergency care should be obtained directly rather than through the CHAMP App.

SUMMARY:
This is a multi-site research study with an optional research repository that will consist of clinically derived data and photographic or video images of patients in the home setting with complex health conditions to evaluate the safety and efficacy of the CHAMP® software platform, with data and photographic or video images input and/or uploaded by the parent or other legally authorized representative (LAR) of patients with complex congenital heart disease as a target population.

DETAILED DESCRIPTION:
Study objectives

1. To evaluate whether data collection and transmission through the CHAMP software platform improves communication between health care providers and parents/LAR that positively affects the care of children with complex congenital heart disease in which asynchronous monitoring in the home setting is indicated
2. To determine the accuracy of data obtained regarding observation by parent or caregiver of the condition of children with complex congenital heart disease in which asynchronous monitoring in the home setting is indicated.
3. To evaluate the use of the CHAMP App for clinical purposes, including user satisfaction with the data entry, parental self-management, and transmission capabilities.
4. To evaluate the real-world performance analytics (RWPA) of the CHAMP software platform for transfer of parent-entered data for children with complex congenital heart disease in which asynchronous monitoring in the home setting is indicated.

Endpoints

1. To demonstrate that parents and caregivers for children with complex congenital heart disease in which asynchronous monitoring in the home setting is indicated can accurately identify and transmit to healthcare providers specific health-related data including intake of food, fluids and mediations; output, including urination, defecation, and vomiting; weight; vital signs including oxygen saturation as measured by pulse oximetry; heart rate as measured either by a heart rate monitor or manually by the parent or caregiver; and temperature, measured by a reliable thermometer; and the value and reliability of videos provided by parents and caregivers regarding behavior of pediatric study participants for use in evaluating participant's health status.
2. To demonstrate that data obtained through the use of devices such as pulse oximeters, as entered into the app by parents and caregivers, provide valuable information regarding the health status of children with Complex Diagnoses in a home setting.
3. To demonstrate characteristics of CHAMP through real world health analytics (RWHA), user experience analytics (UX), and product performance analytics (PPA).

The study duration is open-ended for safety, effectiveness, and performance of the CHAMP app. Unless consent is withdrawn, data will be kept and used for data analysis and, if consented to the research repository for multi-site research purposes indefinitely. At age 18, previously pediatric patients may be approached for reconsent.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-17 years with a parent/Legally authorized representative
* Diagnosed with a complex health condition in which asynchronous monitoring in the home setting is appropriate.
* Pediatric patient's cardiac care team has decided that the patient's treatment plan may benefit from remote home monitoring.
* Institution that the subject is followed through clinically has been an approved as site for the CHAMP app study with Children's Mercy Kansas City.

Adult participants

* Parents/Legally authorized representatives of pediatric subject.
* Healthcare team users at an institution that is an approved site for the CHAMP app Study with Children's Mercy Kansas City.

Exclusion Criteria:

* Inability to be discharged to care in the home setting.
* Those not meeting the above inclusion criteria.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with complex congenital heart disease in which asynchronous monitoring in the home setting is indicated in the home setting through a multi-regional approach.
  Parents who utilize their CHAMP App and the healthcare team that log-in are also part of the CHAMP App study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Human factors/usability engineering: Login failures | Over a 3 month period
  Rate of attempts of log-in failures
Human factors/usability engineering: Imprecision | Over a 3 month period
  Rate of data values reported with imprecision
Clinical Safety: Anticipated adverse events | Over a 3 month period
  Anticipated Adverse event rates
Clinical Safety: Event resolution- anticipated | Time in days, reported over the last 3 months
  Time to resolve anticipated adverse events
Clinical Safety: Unanticipated Adverse events | Time in days, reported over the last 3 months
  Unanticipated adverse event rates
Clinical Safety: Event resolution- unanticipated | Time in days, reported over the last 3 months
  Time to resolve unanticipated adverse events
Health Benefits: Adherence | Measurement of adherence to daily data entry per each patient/parent over 3 month period on non-hospitalized days, during the study period
  Rate of adherence to daily data entry
User Satisfaction: Complaints | Over a 3 month period
  Complaint rates via the healthcare team web portal
User Satisfaction CHAMP Video | through study completion, an average of 9 months
  Feedback from healthcare team will be received via treatment endpoint survey questions. Likert scale questions 1-strongly disagree to 5 strongly agree (Using CHAMP videos for the interstage monitoring of this patient improved clinical decisions for the home monitoring team). Available to put in comments.
User Satisfaction: Communication | through study completion, an average of 9 months
  Feedback from healthcare team will be received via treatment endpoint survey questions Likert scale questions 1-strongly disagree to 5 strongly agree ( Using CHAMP for the interstage monitoring of this patient improved communication with the parents at home.) Available to put in comments.
User Engagement | Over a 3 month perriod
  Total number of registered users (Active, treatment endpoint reached) and data totals per parent entered measure. De-identified Demographics and age areas utilization -Utilization across the number of pediatric sites, healthcare teams
CHAMP app performance: Downtime | Over a 3 month period
  Product Performance Analytics measured through Any system downtime
CHAMP app performance: Cybersecurity | Over a 3 month period
  Product Performance Analytics measured through Any reported breaches
CHAMP app performance | Quarterly review of CHAMP App Performance will be measure over the preceding 3 months for frequency of changes required
  Product Performance Analytics measured through --Bug/defect rate or Version failure rates

CONTACTS AND LOCATIONS:
Overall Officials: Lori Erickson, PhD, Principal Investigator — Director, Remote Health Solutions Children's Mercy
Locations (9):
- United States (9):
  - Children's National Hospital, Washington D.C., District of Columbia
  - Nicklaus Variety Children's Hospital, Miami, Florida
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Cook's Children's, Forth Worth, Texas
  - Children's Memorial Hermann Hospital, Houston, Texas
  - Primary Children's Hospital/University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shirali G, Erickson L, Apperson J, Goggin K, Williams D, Reid K, Bradley-Ewing A, Tucker D, Bingler M, Spertus J, Rabbitt L, Stroup R. Harnessing Teams and Technology to Improve Outcomes in Infants With Single Ventricle. Circ Cardiovasc Qual Outcomes. 2016 May;9(3):303-11. doi: 10.1161/CIRCOUTCOMES.115.002452. Epub 2016 May 10. PMID 27166202
- [Background] Bingler M, Erickson LA, Reid KJ, Lee B, O'Brien J, Apperson J, Goggin K, Shirali G. Interstage Outcomes in Infants With Single Ventricle Heart Disease Comparing Home Monitoring Technology to Three-Ring Binder Documentation: A Randomized Crossover Study. World J Pediatr Congenit Heart Surg. 2018 May;9(3):305-314. doi: 10.1177/2150135118762401. PMID 29692236
- [Background] Aly DM, Erickson LA, Hancock H, Apperson JW, Gaddis M, Shirali G, Goudar S. Ability of Video Telemetry to Predict Unplanned Hospital Admissions for Single Ventricle Infants. J Am Heart Assoc. 2021 Aug 17;10(16):e020851. doi: 10.1161/JAHA.121.020851. Epub 2021 Aug 7. PMID 34365801
- [Background] Erickson LA, Emerson A, Russell CL. Parental mobile health adherence to symptom home monitoring for infants with congenital heart disease during the single ventricle interstage period: A concept analysis. J Spec Pediatr Nurs. 2020 Oct;25(4):e12303. doi: 10.1111/jspn.12303. Epub 2020 Jul 14. PMID 32662243
- [Background] Patel PS, Shah SK, Feldman K, Hancock HS, Moehlmann ML, Ricketts A, Files MD, McFarland C, Erickson L, Romans RA. Associations of Home Monitoring Data to Interventional Catheterization for Infants with Recurrent Coarctation of the Aorta and Hypoplastic Left Heart Syndrome. Pediatr Cardiol. 2023 Oct;44(7):1462-1470. doi: 10.1007/s00246-023-03224-8. Epub 2023 Jul 8. PMID 37421465